CLINICAL TRIAL: NCT03795168
Title: Transcranial Vibrating System for Improving Outcomes of Vestibular Physical Therapy
Brief Title: Transcranial Vibrating System for Improving Vestibular Physical Therapy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study center closed down
Sponsor: Otolith Labs (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: OLith10301
Record Dates: First submitted 2019-01-01; First posted 2019-01-07 (Actual); Last update posted 2022-04-01 (Actual); Status verified 2022-03

CONDITIONS: Vertigo; Dizziness; Nausea; Balance
Keywords: Vestibular physical therapy; Positional vertigo; Ménière's disease
MeSH Terms: conditions — Vertigo; Dizziness; Nausea; Meniere Disease

STUDY DESIGN:
Intervention Model Description: Arm 1: Participants undergoing vestibular physical therapy (PT) will perform PT exercises with or without wearing the transcranial vibrating system (TCVS). Following the end of their PT exercises (30 minutes or less if the participant was too dizzy to finish), participants will evaluate dizziness using a dizziness symptom scale (DSS) and PT exercise duration will be recorded. A force plate system assessment will also be performed with or without wearing the TCVS during the first and last PT visit to evaluate participant's balance.
  Arm 2: Participants will undergo the identical protocol as arm 1 with the exception that participants will wear the TCVS at optimal vibration frequency or the TCVS at irrelevant vibration frequency (sham).
  To determine TCVD's effect on dizziness and balance, the outcomes measured in both arms (1. DSS, 2. duration of PT exercise, 3. balance) will be compared statistically between:
  * TCVD versus no device
  * TCVD optimal frequency versus TCVD sham
Who Masked: Participant, Investigator
Masking Description: Arm 1: their will be no masking as the participants will either wear the transcranial vibrating system (TCVS) or not.
  Arm 2: the investigators will be provided 2 TCVS by the sponsor, labeled A or B, which will be randomly assigned to participants by the sponsor. One TCVS will be set at the optimal vibration frequency and the other TCVS will be set at an irrelevant vibration frequency (sham). The investigators and the participants will not know which TCVS is optimal or sham, thus the arm 2 will be double blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Transcranial vibrating system effect (Experimental): Participants will be enrolled for a 4 week period and will have 2 vestibular physical therapy (PT) visits per week. During the first 2 weeks (4 visits), 20 participants will perform their PT exercises (30 minutes or less if the participant is too dizzy to finish) wearing the transcranial vibration system (TCVS) and the other 20 participants without. The following 2 consecutive weeks (4 visits), participants will perform their PT exercises wearing the TCVS if they weren't previously, or won't wear the device during their PT exercises if they were previously.
  Outcomes measured:
  * at every visit: dizziness at the end of PT exercise (with dizziness symptom scale DSS); duration of PT exercise
  * at the first and last visit: force plate system assessment (balance)
  Interventions: Device: Transcranial vibrating system
- Vs transcranial vibrating system sham (Sham Comparator): 40 participants will be enrolled for a 4 week period and will have 2 vestibular physical therapy (PT) visits per week. Participants will perform their PT exercises (30 minutes or less if the participant is too dizzy to finish) wearing the transcranial vibration system (TCVS) at optimal vibrating frequency or wearing the TCVS at irrelevant vibrating frequency (sham). The TCVS and TCVS sham will be labeled A or B by the sponsor. The investigators and participants will not know which TCVS is optimal or sham. The sponsor will randomly assign participants TCVS A or B.
  Outcomes measured:
  * at every visit: dizziness at the end of PT exercise (with dizziness symptom scale DSS); duration of PT exercise
  * at the first and last visit: force plate system assessment (balance)
  Interventions: Device: Transcranial vibrating system; Device: Transcranial vibrating system sham

INTERVENTIONS:
Device: Transcranial vibrating system — The transcranial vibrating system (TCVS) will be worn by participants performing vestibular physical therapy (PT) exercises. The TCVS vibrating element will be placed against the skull, preferably over the mastoid bone behind the ear and will be hold in place by a headband. The TCVS will be worn during the whole time of the vestibular PT exercise (30 minutes) or less if the participant is unable to complete its exercises. The TCVS will be set at an optimal vibration frequency as determined in a previous study.
Device: Transcranial vibrating system sham — A transcranial vibrating system (TCVS) sham set at an irrelevant vibrating frequency will be worn by participants performing vestibular physical therapy (PT) exercises in arm 2. The TCVS sham vibrating element will be placed against the skull, preferably over the mastoid bone behind the ear and will be hold in place by a headband. The TCVS sham will be worn during the whole time of the vestibular PT exercise (30 minutes) or less if the participant is unable to complete its exercises.
  Arms: Vs transcranial vibrating system sham

SUMMARY:
This research study aims to determine whether low-frequency transcranial vibrations can act as a possible treatment for the dizziness and nausea often associated with vestibular physical therapy.

DETAILED DESCRIPTION:
The purpose of this study is to determine the effectiveness of a Transcranial Vibration System (TCVS) at reducing the increased nausea and discomfort sometimes associated with vestibular physical therapy. The TCVS is a small device attached to an elastic band. It is worn around the head and produces vibrations. There is no implant or surgical procedure. The FDA has made a pre-determination that this is a low-risk device (a "Class 2 device" in FDA terminology).

The TCVS has previously been tested in healthy volunteers and has been found to safely and effectively decrease dizziness and nausea associated with vestibular discomfort. This study will expand that research to vestibular disorder patients who are undergoing physical therapy. The study compares the outcomes to not wearing a device, or to a control (inneffective) device.

ELIGIBILITY:
Inclusion Criteria:

* reluctant or unable to perform a full session of vestibular physical therapy

Exclusion Criteria:

* History of head injury within the last six months or currently suffering the effects of a head injury (i.e. concussion or traumatic brain injury)
* Presence of severe aphasia.
* History of diagnosed neuropsychiatric disorders (e.g. hypochondriasis, major depression, schizophrenia).
* Documented neurodegenerative disorders.
* Pregnancy Female candidates will be asked to take a pregnancy test first and will have to make a informed decision to participate based on the results of the pregnancy test.
* History of Cerebrovascular disorders.
* History of ear operation other than myringotomy and tube placement in the past.
* Systemic disorders to include chronic renal failure, cirrhosis of the liver, autoimmune disease, heart disease, lung disease, or severe arthritis.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
Change in duration of the vestibular physical therapy exercise session | up to 30 minutes
  The participants will perform vestibular physical therapy exercises for 30 minutes unless their dizziness symptoms prevend them to finish. The change in vestibular physical therapy exercises they can perform will be recorded by the investigator. This value will be recorded immediately after they finish their physical therapy exercises.
Change in dizziness index | Questionaire immediately after the end of physical therapy exercise
  The dizziness index will be evaluated with the Dizziness Symptom Scale (DSS) with a scale from 1 (no dizziness) to 10 (strong dizziness). The change of DSS will be evaluated between participants wearing:
  * the transcranial vibrating system (TCVS)
  * no TCVS
  * the TCVS sham
Change in balance | During first and last vestibular physical therapy visit; expected duration maximum 10 minutes
  Participant's balance will be evaluated with a force plate platform (Bertec Device). Participants will be placed on the plate 1. eyes open, 2. eyes closed, 3. eyes open while standing on a foam pad, 4. eyes closed while standing on a foam pad. Each of the 4 conditions will involve the participant standing barefoot on a force plate platform for 10 seconds. The change in participant's balance (X&Y direction) will be assessed by recording values of the Bertec device in two conditions: first with participants not wearing the TCVS and second with participants wearing the TCVS at optimal vibration frequency or wearing the TCVS sham. Clinical parameters obtained from the Bertec system will be recorded, including "falls" and will be compared between conditions to evaluate participant's change in balance. Participants will always be held safe with a harness secured to a mount point in the ceiling.

CONTACTS AND LOCATIONS:
Overall Officials: Didier Depireux, PhD, Study Director — Otolith Labs
Locations (2):
- United States (2):
  - Fyzical - Dizziness and Fall Prevention - Shady Grove, Rockville, Maryland
  - FYZICAL Therapy & Balance Center of Rockville, Rockville, Maryland

IPD SHARING:
Plan to Share IPD: No